CLINICAL TRIAL: NCT05837234
Title: A Prospective, Open-Label, Multi-Center Trial to Evaluate the Safety and Effectiveness of Ultra Low Frequency Spinal Cord Stimulation in Patients With Chronic Low Back Pain
Brief Title: Ultra Low Frequency Spinal Cord Stimulation for Chronic Low Back Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Presidio Medical, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PMH-003
Record Dates: First submitted 2023-04-19; First posted 2023-05-01 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Chronic Pain; Chronic Low-back Pain
Keywords: Neuromodulation; Spinal Cord Stimulation
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- ULF SCS (Experimental): Participants with chronic low back pain that is refractory to conservative care will undergo temporary trial stimulation with the ULF SCS system. Those receiving at least 50% pain relief of their chronic back pain will be eligible for a permanent device implant and followed for 24 months.
  Interventions: Device: ULF SCS

INTERVENTIONS:
Device: ULF SCS — Ultra low frequency spinal cord stimulation

SUMMARY:
The Presidio Medical Ultra Low Frequency (ULF™) Spinal Cord Stimulation (SCS) System is intended to provide pain relief to participants who have been clinically diagnosed with chronic low back pain with or without leg pain.

DETAILED DESCRIPTION:
This is a prospective, open-label, multi-center clinical trial in which participants with chronic low back pain (CLBP) with/without leg pain will be invited to enroll and undergo treatment with the ULF SCS system. The purpose of this study is to evaluate the safety and effectiveness of ULF SCS over a 3-year period.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with chronic low back pain with/without leg pain (VAS ≥60mm for back pain for the past week), which has been refractory to conservative therapy for a minimum of 3 months.
2. Be on no or stable pain medications, as determined by the investigator, for at least 28 days prior to the screening visit.
3. Is currently considered medically stable as judged by investigator.
4. Able to operate the SCS device (e.g., using remote control) and charge the device appropriately.
5. Determined to be a good surgical candidate by the investigator.
6. Willing to sign the Human Research Ethics Committee (HREC) approved informed consent and deemed capable of complying with the requirements of the study protocol.
7. Willing to stay on stable medications until implantable pulse generator (IPG) activation (i.e., from IPG implant to IPG activation, except for usual postoperative medications required following IPG insertion).
8. Able to comply with study requirements and attend all scheduled visits.
9. Eighteen (18) years of age or older.
10. Literate, able to speak English and able to complete questionnaires independently.

Exclusion Criteria:

1. Diagnosis of active disruptive psychological or psychiatric disorder or other known condition significant enough to impact perception of pain, compliance, intervention and/or ability to evaluate treatment outcome as assessed by a clinical psychologist or psychiatrist in a psychological assessment performed at Baseline.
2. Chronic pain in any area other than back or legs, such that it precludes subject's ability to assess their pain for the primary indication of chronic low back pain as determined by Investigator.
3. Previous experience with implantable neuromodulation devices (e.g., spinal cord stimulation, peripheral nerve stimulation, dorsal root ganglion stimulation).
4. Opioid usage with average total daily morphine equivalent dose (MED) of >60 mg.
5. A known need for an MRI or surgery within a 2-week period of the screening visit through the end of the study.
6. Female candidates of childbearing potential that are pregnant (confirmed by positive urine/blood pregnancy test) or plan to get pregnant during the duration of the study.
7. Subject is participating in another interventional clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2023-05-09 (Actual); Primary Completion 2025-05-19 (Actual); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Back pain responder rate at 3 months as assessed using a visual analog scale (VAS) | 3 months
  A responder is defined as a participant that achieved at least 50% reduction in back pain at the follow-up compared to baseline. Responder rate is defined as the percentage of participants that were responders.

SECONDARY OUTCOMES:
Change in back pain VAS at 3 months | 3 months
  The mean percentage change in VAS back pain intensity from baseline.
Change in back pain VAS at 6 months | 6 months
  The mean percentage change in VAS back pain intensity from baseline.
Change in back pain VAS at 12 months | 12 months
  The mean percentage change in VAS back pain intensity from baseline.
Change in leg pain VAS at 3 months | 3 months
  The mean percentage change in VAS leg pain intensity from baseline. Calculated only for participants who scored at least 40 out of 100mm for leg pain at baseline.
Change in leg pain VAS at 6 months | 6 months
  The mean percentage change in VAS leg pain intensity from baseline. Calculated only for participants who scored at least 40 out of 100mm for leg pain at baseline.
Change in leg pain VAS at 12 months | 12 months
  The mean percentage change in VAS leg pain intensity from baseline. Calculated only for participants who scored at least 40 out of 100mm for leg pain at baseline.
Proportion of participants with a minimal clinically important difference (MCID) as measured by Oswestry Disability Index (ODI) at 3 months | 3 months
  The MCID is defined as at least a 10-point improvement on ODI.
Proportion of participants with a MCID as measured by ODI at 6 months | 6 months
  The MCID is defined as at least a 10-point improvement on ODI.
Proportion of participants with a MCID as measured by ODI at 12 months | 12 months
  The MCID is defined as at least a 10-point improvement on ODI.
Change in EuroQol-5 Dimension (EQ-5D) quality of life index at 3 months | 3 months
  The mean change in EQ-5D index from baseline.
Change in EQ-5D quality of life index at 6 months | 6 months
  The mean change in EQ-5D index from baseline.
Change in EQ-5D quality of life index at 12 months | 12 months
  The mean change in EQ-5D index from baseline.
Proportion of participants with remission of low back pain as assessed by VAS at 6 months | 6 months
  Remission is defined as VAS score of 30mm or less for 6 consecutive months.
Proportion of participants with remission of low back pain as assessed by VAS at 9 months | 9 months
  Remission is defined as VAS score of 30mm or less for 6 consecutive months.
Proportion of participants with remission of low back pain as assessed by VAS at 12 months | 12 months
  Remission is defined as VAS score of 30mm or less for 6 consecutive months.
Change in sleep quality as assessed by Medical Outcomes Study Sleep Scale (MOS-SS) at 3 months | 3 months
  The mean change in MOS-SS index from baseline.
Change in sleep quality as assessed by MOS-SS at 6 months | 6 months
  The mean change in MOS-SS index from baseline.
Change in sleep quality as assessed by MOS-SS at 12 months | 12 months
  The mean change in MOS-SS index from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Willem Volschenk, MBCHB, Principal Investigator — Genesis Research Services; Mattew Green, BMBS, Principal Investigator — CerCare; Paul Verrills, MBBS, Principal Investigator — Monash House Research Centre
Locations (3):
- Australia (3):
  - Genesis Research Services Pty Ltd, Newcastle, New South Wales
  - CerCare Pty Ltd, Wayville, South Australia
  - Monash House Research Centre, Clayton, Victoria

IPD SHARING:
Plan to Share IPD: No